CLINICAL TRIAL: NCT04733287
Title: Improving Critical Power and Muscle Function in Older Adults With Heat Therapy
Brief Title: Heat Therapy and Muscle Function Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brigham Young University (Other)
Responsible Party: Principal Investigator, Jayson Gifford, Assistant Professor, Brigham Young University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F2020-023
Record Dates: First submitted 2020-10-14; First posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Exercise Intolerance; Aging; Heat Therapy; High Intensity Interval Training
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Intervention Model Description: Young (18-35 years) and Older (60+ years) will be randomly assigned to one of 3 different conditions (High Intensity Exercise Training of the Knee Extensors, Heat therapy of the Knee Extensors or Sham Heat therapy of the Knee Extensors). Muscle function will be measured before and after 6 weeks of the randomized treatment.
  A separate set of 40 young adults (18-35 years) will undergo 2 weeks of leg immobilization. Half of the subjects will receive daily heat therapy, while the other half will receive a sham heat therapy treatment. Muscle function and critical power will be measured before and after immobilization for both groups
Who Masked: Participant
Masking Description: Subjects assigned to the heat therapy and the sham heat therapy will not know if they are truly receiving the heat therapy or not. The muscle heater (shortwave diathermy) will be placed on the muscle during each visit, but, unbeknownst to the heat and sham group, will not be turned on for the sham group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Effect of High Intensity Interval Training (Experimental): Young and older subjects will participate in single-leg, high-intensity interval training of the right knee extensors (4 intervals of 4 minutes at 80% of max aerobic power with 4 minute rest intervals between, 3x per week for 6 weeks).
  Muscle function and knee extensor critical power will be measured before and after the 6 weeks of treatment.
  Interventions: Other: High Intensity Interval Training of the Knee Extensors
- Effect of Muscle Heat Therapy (Experimental): Young and older subjects will participate in single-leg,heat therapy training of a single leg ( quadriceps femoris, 120 minutes of shortwave diathermy to raise the muscle temperature to ~39C) 3 times a week for 6 weeks.
  Muscle function and knee extensor critical power will be measured before and after the 6 weeks of treatment.
  Interventions: Other: Muscle Heat Therapy
- Effect of Sham Muscle Heat Therapy (Sham Comparator): Young and older subjects will participate in a sham treatment of single-leg,heat therapy training of the right knee extensors (120 minutes with shortwave diathermy unit positioned on leg, but not turned on) 3 times a week for 6 weeks.
  Muscle function and knee extensor critical power will be measured before and after the 6 weeks of treatment.
  Interventions: Other: Sham Heat Therapy
- Effect of Immobilization with Daily Sham Heat Therapy (Sham Comparator): Young subjects (18-35 years) will undergo 2 weeks of leg immobilization while receiving 2 hours of a sham heat therapy treatment each day. For the sham treatment, the heating device will be applied to the limb, but, unbeknownst to the participant, it will not be turned on.
  Muscle function and knee extensor critical power will be measured before and after the 2 weeks of leg immobilization.
  Interventions: Other: Sham Heat Therapy
- Effect of Immobilization with Daily Heat Therapy (Experimental): Young subjects (18-35 years) will undergo 2 weeks of leg immobilization while receiving 2 hours of heat therapy treatment each day. Heat therapy will consist of 120 minutes of shortwave diathermy to raise the quadriceps femoris muscle temperature to ~39C.
  Muscle function and knee extensor critical power will be measured before and after the 2 weeks of leg immobilization.
  Interventions: Other: Muscle Disuse

INTERVENTIONS:
Other: High Intensity Interval Training of the Knee Extensors — Subjects will perform intense, single leg knee extension exercise 3 times a week for 6 weeks. Specifically, subjects will be seated in a custom knee extension ergometer and perform single leg, dynamic knee extension (similar to single leg cycling) as they perform the exercise. After a 6 minute warm-up at ~20% of that leg's maximum aerobic power (determined during a graded exercise test of single leg knee extension), subjects will perform 4 bouts of 4 minutes at ~80% of maximum aerobic power. Recovery of 4 minutes at ~40% will occur between each bout of exercise. A cool down will be provided at the end of exercise. In total, subjects will perform 40 minutes of single leg knee extension exercise, 3 times a week for 6 weeks.
  Maximum aerobic power (determined by a graded exercise test) will be determined again at 3 weeks to appropriately adjust the training intensity.
  Other Names: HIIT
  Arms: Effect of High Intensity Interval Training
Other: Muscle Heat Therapy — Subjects will receive muscle heat therapy on the knee extensor muscles (short-wave diathermy) for 120 minutes for each visit. Specifically, subjects will lie supine while short-wave diathermy units (Megapulse II) will be placed on the quadriceps femoris and turned on to 800 pulses per second with a pulse duration of 400 microseconds. Our previous research (e.g. Hafen et al 2018- Repeated exposure to heat stress...) has indicated that this treatment raises muscle temperature to ~39C, a similar temperature induced by exercise.
  Other Names: Short-wave Diathermy
  Arms: Effect of Muscle Heat Therapy
Other: Muscle Disuse — Subjects will undergo 2 weeks of limb immobilization (a model of muscle disuse). Specifically, a knee brace will be placed on one of the subjects' legs and bent to a flexion of 60 degrees to prevent the foot from touching the ground while standing. Subjects will given a pair of crutches and asked to ambulate on crutches for 2 weeks, avoiding bearing any weight with the immobilized leg.
  Other Names: Leg Immobilization
  Arms: Effect of Immobilization with Daily Heat Therapy
Other: Sham Heat Therapy — Specifically, subjects randomly assigned to the sham group will receive the same treatment as the heat group (same number of visits and set up with the heating units applied to leg for 2 hours each visit) except, unbeknownst to either group, the heating units will never be turned on for the sham group.
  Arms: Effect of Immobilization with Daily Sham Heat Therapy; Effect of Sham Muscle Heat Therapy

SUMMARY:
Exercise tolerance decreases with age and a sedentary lifestyle. Muscle critical power (CP), is a sensitive measure of exercise tolerance that is more even more relevant to and predictive of endurance performance than VO2max.

While recent evidence indicates that CP and muscle function decrease with aging, the cause of this decrease in CP and the best way to mitigate the decrease in CP are unknown.

This study will:

1. Measure knee extensor CP in young and old individuals and determine the extent to which changes in muscle oxygen delivery (e.g. resistance artery function, maximum exercise blood flow), muscle mass and composition (e.g. whole-muscle size, muscle fiber cross-sectional area) and mitochondrial oxygen consumption (e.g. maximal coupled respiration of permeabilized fibers biopsied from the knee extensors) contribute to the decrease in CP with age.
2. Examine the effectiveness of two different therapies (1. High Intensity Interval Training, HIIT and 2. Muscle Heat Therapy) at improving muscle function and critical power in young and older adults.
3. Examine the impact of muscle disuse (2 weeks of leg immobilization), a potential contributor to the decrease in muscle function with aging, on muscle function and critical power and determine if heat therapy is an effective means of minimizing the impact of disuse on muscle function and critical power.

ELIGIBILITY:
Inclusion Criteria:

* 18-95 years of age
* Currently no cardiovascular or metabolic disease (e.g. heart failure, diabetes)
* ability to perform knee extension exercise

Exclusion Criteria:

* Pregnant
* Current cardiovascular or metabolic disease (e.g. heart failure, diabetes)
* participating in exercise training within the last 6 months
* inability to perform knee extension exercise

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Critical Power | 3-8 weeks
  Muscle exercise tolerance, quantified as critical power, will be assessed before and after each intervention. The main outcome will be the change in critical power, expressed in Watts, elicited by each intervention.
  Specifically, participants will perform 3-5 different power outputs of single leg knee extension exercise as long as they can. Subsequently, the line of best fit between the total work performed and duration of each power output trial will be used to quantify critical power, expressed in Watts.

SECONDARY OUTCOMES:
Resistance Artery Function | 3-8 weeks
  Resistance Artery Function will be assessed with the Passive Leg Movement (PLM) technique before and after each intervention. The main variable of interest will be the change in peak blood flow elicited by PLM from before to after each intervention.
  Specifically, PLM will be performed with a member of the research team moving a subject's knee joint through a 90 degree range of motion, at a rate of 1 Hz for 60 seconds. This passive movement elicits a hyperemic response that will will be quantified with Doppler ultrasound of the femoral artery and expressed in ml/min. The highest 1-second average of blood flow to occur during the movement will be identified as the peak blood flow response.
  The main variable of interest will be the change in peak blood flow elicited by PLM from before to after each intervention.
Maximum Exercise Blood Flow | 3-8 weeks
  The maximum rate of blood flow achieved during exercise will be determined before and after each intervention. The main variable of interest will be the change in maximum exercise blood flow from before to after each intervention, expressed in ml/min.
  Specifically, exercise blood flow will be assessed by quantifying the peak hyperemic response, expressed in ml/min, to active single leg knee extension exercise. Following a warm-up, subjects will perform maximal single leg knee extension exercise for 3 minutes while blood flow is quantified with Doppler ultrasound (Logiq E, GE) of the femoral artery. The average rate of blood flow achieved during the final 30 seconds of the exercise will be identified as the maximum exercise blood flow, expressed in ml/min.
Muscle Fiber Size | 3-8 weeks
  The cross-sectional area of muscle fibers biopsied from the treated vastus lateralis will be used to quantify the size of muscle size before and after each intervention. The main variable of interest will be the change in average myofiber cross-sectional area, expressed in square micrometers, from before to after each intervention.
  Specifically, muscle biopsy samples will be mounted on a cork in tragacanth gum . Frozen samples will be adhered to a microscope slide for staining. Slides will be incubated with fluorescently labeled antibodies. CSA will be quantified for each fiber using Olympus CellSens software and subsequently averaged for all fibers on the slide.
Muscle Mitochondrial Function | 3-8 weeks
  Muscle mitochondrial function will be measured in permeabilized fibers biopsied from the vastus lateralis before and after each intervention.
  Specifically, maximal coupled respiration (i.e. OXPHOS or State 3) will be measured with a clark-type electrode (O2K, Oroboros) and expressed in picomoles of oxygen consumed per second.
  The main variable of interest will be the change in Maximal Couple Respiration from before to after each intervention.
Vastus Lateralis Cross-Sectional Area | 3-8 weeks
  The cross-sectional area of the treated vastus lateralis will be measured with magnetic resonance imaging before and after each intervention. The main variable of interest will be the change in cross-sectional area, expressed in square centimeters, from before to after each intervention.
  Specifically, MRI will be used to assess whole muscle cross sectional area of the vastus lateralis. Participants will be scanned while laying supine in a 3.0 Tesla MRI scanner (Siemens). A stock Siemens 2-D multi-slice gradient-recalled echo (GRE) MRI pulse sequence will be used. Images will be takin in slices every 5mm, resulting in a total sequence time of approximately 2-min. This will provide cross-sectional images of the vastus lateralis from the base of the femur (distal condyles) up to the groin. .

CONTACTS AND LOCATIONS:
Overall Officials: Jayson Gifford, Ph.D., Study Director — Brigham Young University; Robert Hyldahl, Ph.D., Principal Investigator — Brigham Young Univeristy
Locations (1):
- Brigham Young University, Provo, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gifford JR, Richardson RS. CORP: Ultrasound assessment of vascular function with the passive leg movement technique. J Appl Physiol (1985). 2017 Dec 1;123(6):1708-1720. doi: 10.1152/japplphysiol.00557.2017. Epub 2017 Sep 7. PMID 28883048
- [Background] Park SY, Ives SJ, Gifford JR, Andtbacka RH, Hyngstrom JR, Reese V, Layec G, Bharath LP, Symons JD, Richardson RS. Impact of age on the vasodilatory function of human skeletal muscle feed arteries. Am J Physiol Heart Circ Physiol. 2016 Jan 15;310(2):H217-25. doi: 10.1152/ajpheart.00716.2015. Epub 2015 Nov 20. PMID 26589330
- [Background] Gifford JR, Garten RS, Nelson AD, Trinity JD, Layec G, Witman MA, Weavil JC, Mangum T, Hart C, Etheredge C, Jessop J, Bledsoe A, Morgan DE, Wray DW, Rossman MJ, Richardson RS. Symmorphosis and skeletal muscle V̇O2 max : in vivo and in vitro measures reveal differing constraints in the exercise-trained and untrained human. J Physiol. 2016 Mar 15;594(6):1741-51. doi: 10.1113/JP271229. Epub 2016 Jan 19. PMID 26614395
- [Background] Hanson BE, Proffit M, Gifford JR. Vascular function is related to blood flow during high-intensity, but not low-intensity, knee extension exercise. J Appl Physiol (1985). 2020 Mar 1;128(3):698-708. doi: 10.1152/japplphysiol.00671.2019. Epub 2020 Jan 9. PMID 31917628
- [Background] Hafen PS, Preece CN, Sorensen JR, Hancock CR, Hyldahl RD. Repeated exposure to heat stress induces mitochondrial adaptation in human skeletal muscle. J Appl Physiol (1985). 2018 Nov 1;125(5):1447-1455. doi: 10.1152/japplphysiol.00383.2018. Epub 2018 Jul 19. PMID 30024339
- [Background] Hafen PS, Abbott K, Bowden J, Lopiano R, Hancock CR, Hyldahl RD. Daily heat treatment maintains mitochondrial function and attenuates atrophy in human skeletal muscle subjected to immobilization. J Appl Physiol (1985). 2019 Jul 1;127(1):47-57. doi: 10.1152/japplphysiol.01098.2018. Epub 2019 May 2. PMID 31046520
- [Background] Poole DC, Burnley M, Vanhatalo A, Rossiter HB, Jones AM. Critical Power: An Important Fatigue Threshold in Exercise Physiology. Med Sci Sports Exerc. 2016 Nov;48(11):2320-2334. doi: 10.1249/MSS.0000000000000939. PMID 27031742
- [Background] Helgerud J, Hoydal K, Wang E, Karlsen T, Berg P, Bjerkaas M, Simonsen T, Helgesen C, Hjorth N, Bach R, Hoff J. Aerobic high-intensity intervals improve VO2max more than moderate training. Med Sci Sports Exerc. 2007 Apr;39(4):665-71. doi: 10.1249/mss.0b013e3180304570. PMID 17414804
- [Background] Brunt VE, Howard MJ, Francisco MA, Ely BR, Minson CT. Passive heat therapy improves endothelial function, arterial stiffness and blood pressure in sedentary humans. J Physiol. 2016 Sep 15;594(18):5329-42. doi: 10.1113/JP272453. Epub 2016 Jun 30. PMID 27270841
- [Background] Kim K, Reid BA, Casey CA, Bender BE, Ro B, Song Q, Trewin AJ, Petersen AC, Kuang S, Gavin TP, Roseguini BT. Effects of repeated local heat therapy on skeletal muscle structure and function in humans. J Appl Physiol (1985). 2020 Mar 1;128(3):483-492. doi: 10.1152/japplphysiol.00701.2019. Epub 2020 Jan 23. PMID 31971474